CLINICAL TRIAL: NCT06532695
Title: Development, ADL, Participation, and Quality of Life in Preterm Infants: Longitudinal Research
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PIFU-CGMH 2023
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-05

CONDITIONS: Preterm Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm: 150 premature infants aged 0-3 years will be collected.
  Interventions: Other: No intervention will be provided.
- Fullterm group: 60 full-term children aged 0-3 years will be collected.
  Interventions: Other: No intervention will be provided.

INTERVENTIONS:
Other: No intervention will be provided. — no intervention will be provided.

SUMMARY:
The three fundamental goals of early rehabilitation for preterm infant after leaving NICU are: optimizing function within each child's prognostic potential, preventing the development of secondary conditions that impact life-long health, and promoting children's participation and qualities in their lives. Understanding knowledges of these developmental patterns of Function and Participation in Life Activities (FPLA) and HRQOL may be helpful for anticipating and managing the problems. This study hypothesizes that the course of developmental patterns in FPLA and HRQOL of preterm infant evolve with their age. The functional recovery levels include developmental function, health, activity, participation, and quality of life (QOL).

Since the previous plan only passed one year and encountered the COVID-19, the number of cases was not as expected. Therefore, this study will use the previous plan to test the functions of reliability, validity, and the evaluation of daily life participation to investigate the long-term performance of premature infants. Vertical development model under tracking. In addition, it is also expected to identify predictors related to the prognosis of preterm infants and compared with the healthy children of the Taiwan Early Childhood Development Survey Database (KIT) to find out the key differences in the developmental function and health of premature infants and healthy children. This study is a three-year longitudinal study of premature infants. It was carried out for three years. 60 full-term children aged 0-3 years and 150 premature infants aged 0-3 years were collected. A total of 210 children underwent a three-year period study. During the follow-up period, in addition to the initial evaluation, each subject will be followed up at 3 months, 6 months, 12 months, 18 months, and 24 months, toddlers( >24months) will be followed up once a year according to the age of KIT's admission, and we will provide caregiver assessment report. We believe the results of this study will improve and support services provided to preterm infants.

DETAILED DESCRIPTION:
Preterm Infant is defined as a group of patients whose gestational age is lower than 37 weeks due to either iatrogenic reasons or maternal reasons. Preterm infant could be classified into 4 group according to gestational age: very early preterm infant, early preterm infant, midterm preterm infant, and late preterm infant. Moreover, they could be categorized into 3 groups of birth weight: extremely low birth weight, very low birth weight, and low birth weight. These varies of preterm infant are indicated to have further developmental and body-functional difficulties and lags. Under the basis of International Classification of Functioning, Disability and Health-Children and Youth Version (ICF-CY) framework, problems related to Preterm infant would further limit their activities of daily living (ADL), participation, and health related quality of life (HRQOL).

The three fundamental goals of early rehabilitation for preterm infant after leaving NICU are: optimizing function within each child's prognostic potential, preventing the development of secondary conditions that impact life-long health, and promoting children's participation and qualities in their lives. Understanding knowledges of these developmental patterns of Function and Participation in Life Activities (FPLA) and HRQOL may be helpful for anticipating and managing the problems. This study hypothesizes that the course of developmental patterns in FPLA and HRQOL of preterm infant evolve with their age. The functional recovery levels include developmental function, health, activity, participation, and quality of life (QOL).

Since the previous plan only passed one year and encountered the COVID-19, the number of cases was not as expected. Therefore, this study will use the previous plan to test the functions of reliability, validity, and the evaluation of daily life participation to investigate the long-term performance of premature infants. Vertical development model under tracking. In addition, it is also expected to identify predictors related to the prognosis of preterm infants and compared with the healthy children of the Taiwan Early Childhood Development Survey Database (KIT) to find out the key differences in the developmental function and health of premature infants and healthy children. This study is a three-year longitudinal study of premature infants. It was carried out for three years. 60 full-term children aged 0-3 years and 150 premature infants aged 0-3 years were collected. A total of 210 children underwent a three-year period study. During the follow-up period, in addition to the initial evaluation, each subject will be followed up at 3 months, 6 months, 12 months, 18 months, and 24 months, toddlers( >24months) will be followed up once a year according to the age of KIT's admission, and we will provide caregiver assessment report. We believe the results of this study will improve and support services provided to preterm infants.

ELIGIBILITY:
Inclusion Criteria:

1. infants with less than 37 weeks of gestation。
2. aged 0-3 years old。
3. caregivers agree and cooperate
4. stable health condition -

Exclusion Criteria:

1. acute health conditions such as infection
2. caregivers or parents cannot communicate in Madarine Chinese.-

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 150 preterm children and 60 fullterm children
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Bayley scales of infant and Toddler Development-fourth edition, Bailey-IV | initial assessemnt, 3 months, 6 months, 12 months, 18 months, and 24 months follow-up
  evaluate the intellegent quatient of the participants
Comprehensive Development Inventory for Infant and Toddlers, CDIIT | initial assessemnt, 3 months, 6 months, 12 months, 18 months, and 24 months follow-up
  evaluate the development of the participants
KIT development and health questionnaire | initial assessemnt, 3 months, 6 months, 12 months, 18 months, and 24 months follow-up
  assess the development and health conditions of the participants
General Movements Assessment, GMA | initial assessemnt, 3 months, 6 months, 12 months, 18 months, and 24 months follow-up
  assess the general movement of the participants
PREMature Infant Index, PREMII | initial assessemnt, 3 months, 6 months, 12 months, 18 months, and 24 months follow-up
  assess the level of premature status

CONTACTS AND LOCATIONS:
Overall Officials: ChiaLing Chen, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No